CLINICAL TRIAL: NCT00001880
Title: Exploratory Study of Non-Myeloablative Allogeneic Stem Cell Transplantation and Donor Lymphocyte Infusions for Metastatic Neoplasms Refractory to Standard Therapy
Brief Title: Stem Cell Transplantation for Metastatic Solid Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was closed early due to lack of accrual
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 990064; 99-H-0064; NCT00003839 (obsolete NCT alias)
Record Dates: First submitted 2006-07-03; First posted 1999-11-04 (Estimated); Results first posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2020-08

CONDITIONS: Neoplasm Metastasis
Keywords: Engraftment; Peripheral Blood Stem Cells; Non-Myeloablative Bone Marrow Transplantation; Metastatic Solid Tumors; Graft-Versus-Host Disease; Cancer; Tumor
MeSH Terms: conditions — Neoplasm Metastasis; Graft vs Host Disease; Neoplasms | interventions — Methotrexate; Cyclosporine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Stem Cell Transplantation in Patients With Progressive and Incurable Metastatic Solid Tumors (Experimental): Cyclosporin beginning day -4 then stem cells given on Day 0 followed by intravenous Methotrexate on days +1, +3, and +6.
  Interventions: Drug: methotrexate; Drug: Cyclosporin

INTERVENTIONS:
Drug: methotrexate — Cyclosporin beginning day -4 and intravenous Methotrexate on days +1, +3, and +6 will be given
  Other Names: MTX (methotrexate)
Drug: Cyclosporin — Cyclosporin beginning day -4 and intravenous Methotrexate on days +1, +3, and +6 will be given
  Other Names: CsA (Cyclosporin)

SUMMARY:
The goal of this research study is to identify other types of cancer (malignant neoplasms) that may be treatable with stem cell transplantation (allogenic peripheral blood stem cell transplantation.

Patients with a variety of different types of cancerous tumors that have spread (metastasized) and whose conditions have not improved with stand therapy, will be eligible to participate. Those patients selected to participate in the study will undergo a procedure known as a "mini-transplant". The mini-transplant is a transplantation of stem-cells collected from a sibling (brother or sister) of the patient. Unlike traditional bone marrow transplants, the mini-transplant does not require intense chemotherapy or radiation therapy. Because of this, patients experience fewer and less severe side effects.

This study is open to patients diagnosed with a variety of metastatic solid tumors including esophageal, gastric (stomach), colon, rectal, liver tumors (hepatoma), cancer of the biliary system (cholangiocarcinoma), cancer of the pancreas, lung, breast, prostate, bone (sarcoma), adrenal basal cell, bladder, and adenocarcinomas of unk primary origin.

DETAILED DESCRIPTION:
The main objective of this study is to identify metastatic neoplasms, which may be susceptible to the GVT effect. We will treat patients with progressive metastatic solid tumors refractory to standard therapy with a non-myeloablative allogeneic PBSC transplant from a family donor. A GVT effect from immunocompetent donor immune cells could extend life expectancy and possibly cure such patients.

Eligible patients will be treated with an allogeneic peripheral blood stem cell transplant from an HLA identical or single HLA antigen-mismatched family donor, using an intensive immunosuppressive regimen without myeloablation ("mini-transplant") in an attempt to decrease the transplant related toxicities while preserving the anti-malignancy and/or anti-host marrow effect of the graft. The low intensity non-myeloablative conditioning regimen should provide adequate immunosuppression to allow stem cell and lymphocyte engraftment. A T-cell replete, donor-derived, granulocyte colony stimulating factor (G-CSF)-mobilized peripheral blood stem cells (PBSC) will be used to establish hematopoietic and lymphoid reconstitution. We will infuse lymphocytes in patients with <100% donor T-cell chimerism or with evidence of tumor progression in an attempt to prevent graft rejection and enhance a graft-versus-malignancy effect, respectively.

This trial is open to several different types of metastatic, treatment-refractory, solid neoplasms, breast, cholangiocarcinoma, small intestine/colon/rectal adenocarcinoma, esophageal/gastric, hepatocellular, pancreatic, prostate, and bony/soft tissue sarcomas. The trial design permits up to 10 patients with a specific tumor type to be enrolled to screen for anti-tumor effects. A single complete response in a specific tumor type is an indication to exclude further patients with that diagnosis from the study. Subsequently, a new protocol which focuses on further defining a GVT effect in that disease category will be instituted.

ELIGIBILITY:
* INCLUSION CRITERIA:

PATIENTS:

Patients with metastatic solid tumors ( breast, cholangiocarcinoma, small intestine/colon/rectal, adenocarcinoma, esophageal/gastric, hepatocellular, pancreatic, prostate, bony/soft tissue sarcomas, which are histologically confirmed, progressive and incurable.

Due to low accrual, effective 12/19/2006, patients with adrenal, basal cell, transitional cell carcinoma of the bladder or uroepithelium, ovarian, small cell lung cancer, non small cell lung cancer, and adenocarcinomas of unknown primary origin are no longer eligible for the trial.

Age greater than or equal to 10 to less than or equal to 80.

No known standard therapy for the patient's disease that is potentially curative or definitely capable of extending life expectancy.

Metastatic disease, which is bi-dimensionally evaluable radiographically.

No prior treatment for neoplasm within 30 days.

Ability to comprehend the investigational nature of the study and provide informed consent.

Availability of HLA identical or single HLA-locus mismatched family donor.

Willingness and availability to return to the NIH for scheduled follow-ups.

DONOR:

HLA identical or single HLA-locus mismatched family donor

Age greater than or equal to 10 up to 80 years old.

Ability to comprehend the investigational nature of the study and provide informed consent.

EXCLUSION CRITERIA:

PATIENT:

Pregnant or lactating.

Age less than 10 or greater than 80 years.

ECOG performance status of 3 or more.

Psychiatric disorder or mental deficiency severe as to make compliance with the BMT treatment unlikely, and making informed consent impossible.

Major anticipated illness or organ failure incompatible with survival from PBSC transplant.

DLCO: less than 40% predicted.

Left ventricular ejection fraction: less than 30%.

Serum creatinine greater than 2.5mg/dl or creatinine clearance less than 50 cc/min by 24 hr urine collection.

Serum bilirubin greater than 4 mg/dl

Transaminases greater than 5 times the upper limit of normal.

Oral intake less than 1,200 calories/day.

Recent weight loss of greater than or equal to 10% of actual body weight.

Life expectancy less than 3 months

Therapy for malignancy within 4 weeks of beginning protocol.

CNS metastatic disease associated with intracranial bleeding, uncontrolled seizure disorder or significant intracranial mass effect.

Other malignant diseases liable to relapse or progress within 5 years.

Uncontrolled infection.

DONOR:

Pregnant or lactating.

Donor unfit to receive G-CSF and undergo apheresis. (Uncontrolled hypertension, history of congestive heart failure or unstable angina, thrombocytopenia).

Age less than 10 or greater than 80 years.

HIV positive. Donors who are positive for HBV, HCV or HTLV-I may be used at the discretion of the investigator following counseling and approval from the recipient.

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 1999-03-12 (Actual); Primary Completion 2008-08-14 (Actual); Study Completion 2020-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Childs, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Eibl B, Schwaighofer H, Nachbaur D, Marth C, Gachter A, Knapp R, Bock G, Gassner C, Schiller L, Petersen F, Niederwieser D. Evidence for a graft-versus-tumor effect in a patient treated with marrow ablative chemotherapy and allogeneic bone marrow transplantation for breast cancer. Blood. 1996 Aug 15;88(4):1501-8. PMID 8695872
- [Background] Or R, Ackerstein A, Nagler A, Kapelushnik J, Naparstek E, Samuel S, Amar A, Bruatbar C, Slavin S. Allogeneic cell-mediated immunotherapy for breast cancer after autologous stem cell transplantation: a clinical pilot study. Cytokines Cell Mol Ther. 1998 Mar;4(1):1-6. PMID 9557210
- [Background] Ueno NT, Rondon G, Mirza NQ, Geisler DK, Anderlini P, Giralt SA, Andersson BS, Claxton DF, Gajewski JL, Khouri IF, Korbling M, Mehra RC, Przepiorka D, Rahman Z, Samuels BI, van Besien K, Hortobagyi GN, Champlin RE. Allogeneic peripheral-blood progenitor-cell transplantation for poor-risk patients with metastatic breast cancer. J Clin Oncol. 1998 Mar;16(3):986-93. doi: 10.1200/JCO.1998.16.3.986. PMID 9508181
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1999-H-0064.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was closed early due to lack of accrual
Groups:
- Stem Cell Transplantation in Patients With Progressive and Incurable Metastatic Solid Tumors: CSA beginning day -4 and intravenous MTX on days +1, +3, and +6 will be given
  methotrexate: CSA beginning day -4 and intravenous MTX on days +1, +3, and +6 will be given
  cyclosporin: CSA beginning day -4 and intravenous MTX on days +1, +3, and +6 will be given
Period: Overall Study
Arm/Group | Stem Cell Transplantation in Patients With Progressive and Incurable Metastatic Solid Tumors
Started | 42
Completed | 28
Not Completed | 14
Not completed — Death | 14

BASELINE CHARACTERISTICS:
Arm/Group | Stem Cell Transplantation in Patients With Progressive and Incurable Metastatic Solid Tumors
Number analyzed (Participants) | 42
Age, Continuous [Median (Full Range); unit: years] — Population: 22 male participants and 20 female participants for total of 42 participants
  years
    Male: number analyzed (Participants) | 22
    Male | 55 [24 to 67]
    Female: number analyzed (Participants) | 20
    Female | 45 [28 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 37
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Based on Tumor Response Criteria With Anti-tumor Effect Induce by Graft-versus-tumor Effect.
Description: To identify an anti-tumor effect of allogenic PNSC transplantation by induction of a graft-versus-tumor (GVT) effect in patients with a diversity of metastatic solid tumors, which are refractory to standard therapy.
  Tumor response assessed as follows:
  Complete response (CR): disappearance of all signs and symptoms of metastatic disease for a period of at least one month.
  Partial response (PR): a 50% or greater decrease in the sum of the products of the longest perpendicular diameters of all measured lesions lasting for a period of at least one month. No new metastatic lesions may appear.
  Stable disease (SD): tumor measurements not meeting the criteria of CR, PR, or PD.
  Progressive disease (PD): increase of 25% or greater in the sum of the products of the longest perpendicular diameters of all measured lesions compared to the smallest previous measurements, or the development of any new metastatic disease.
Time Frame: one year
Measure: Count of Participants; unit: Participants
Arm/Group | Stem Cell Transplantation in Patients With Progressive and Incurable Metastatic Solid Tumors
Number analyzed (Participants) | 42
Participants
  Complete response (CR) | 0
  Partial response (PR) | 9
  Stable disease (SD): | 5
  Progressive disease (PD) | 28

2. Secondary Outcome: Number of Participants That Achieved Engraftment
Description: Number of participants that achieved engraftment based on blood Chimerism Cluster of differentiation 3 (CD3) analysis that is greater than or equal to 95%.
Time Frame: Day 100
Population: 9 participants data was not evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Stem Cell Transplantation in Patients With Progressive and Incurable Metastatic Solid Tumors
Number analyzed (Participants) | 33
Participants | 31

3. Secondary Outcome: Number of Participants Who Received Donor Lymphocyte Infusion to Achieve Tumor Regression or Prevent Graft Failure
Description: To evaluate the effects of donor lymphocyte infusion (DLI) and cyclosporine A (CSA) withdrawal on tumor regression in participants who show progressive disease off of CSA and in the absence of grade > II GVHD, or who are at risk for graft failure due to incomplete donor T-cell engraftment will receive one or more DLI.
  Tumor response assessed as follows:
  Complete response (CR): disappearance of signs & symptoms of metastatic disease at least one month.
  Partial response (PR): a 50% or greater decrease in the sum of the products of the longest perpendicular diameters of all measured lesions lasting at least one month. No new metastatic lesions may appear.
  Stable disease (SD): tumor measurements not meeting the criteria of CR, PR, or PD.
  Progressive disease (PD): increase of 25% or greater in the sum of the products of the longest perpendicular diameters of all measured lesions compared to the smallest previous measurements, or development of new metastatic disease.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Stem Cell Transplantation in Patients With Progressive and Incurable Metastatic Solid Tumors
Number analyzed (Participants) | 42
Participants | 16

4. Secondary Outcome: Number of Participants Who Developed Acute GVHD Grade 2 and Higher
Description: Number of participants who developed Acute Graft vs Host Disease (GVHD) Grades I, II, III, IV as defined by CIMBTR criteria for Organ Stages of Acute GVHD.
  Grades are defined as:
  Grade I: Skin = Maculopapular rash< 25% of body surface area (BSA); Liver = Total Bilirubin 2-3 mg/dL; Lower GI = stool output/day is 500-999 mL/day.
  Grade II: Skin = rash on 25-50 percent body surface area; Liver = Total Bilirubin 3.1-6.0 mg/dL; Lower GI = Diarrhea 1001-1500 mL/day.
  Grade III: Skin = Rash on >50% of body surface; Liver = Total Bilirubin 6.1 - 15.0 mg/dL; Lower GI = Diarrhea > 1500 mL/day.
  Grade IV: Skin = Generalized erythroderma plus bullous formation; Liver = Total Bilirubin >15 mg/dL; Lower GI = Severe abdominal pain with or without ileus.
  Grade I GVHD is characterized as mild disease, grade II GVHD as moderate, grade III as severe, and grade IV life-threatening.
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Stem Cell Transplantation in Patients With Progressive and Incurable Metastatic Solid Tumors
Number analyzed (Participants) | 42
Participants
  Grade II | 9
  Grade III-IV | 11
  No Acute GVHD | 22

5. Secondary Outcome: Number of Participants Who Developed Chronic GVHD
Description: Number of participants who developed Chronic Graft vs Host Disease (GVHD).
  Chronic GVHD is defined as symptoms that persist or appear after 100 days since the time of stem cell transplantation.
Time Frame: Day 100 to year 2
Population: 1 participant passed away prior to day 100 therefore is not evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Stem Cell Transplantation in Patients With Progressive and Incurable Metastatic Solid Tumors
Number analyzed (Participants) | 41
Participants | 18

ADVERSE EVENTS:
Time Frame: 8.5 years
Arm/Group | Stem Cell Transplantation in Patients With Progressive and Incurable Metastatic Solid Tumors
All-Cause Mortality (participants affected / at risk) | 14/42
Serious Adverse Events (participants affected / at risk) | 21/42
Other Adverse Events (participants affected / at risk) | 7/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stem Cell Transplantation in Patients With Progressive and Incurable Metastatic Solid Tumors (N=42)
Mucositis with fever (Gastrointestinal disorders) | 2 (2)
Pseudomonas sepsis (Infections and infestations) | 1 (1)
Parainfluenza pneumonia and septic shock (Infections and infestations) | 1 (1)
Pulmonary aspergillus (Infections and infestations) | 1 (1)
Dyspnea with progressive mets to lungs (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fecal impaction (Gastrointestinal disorders) | 1 (1)
Community acquired pneumonia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (12)
Acute Graft VS Host Disease of GI Tract (Gastrointestinal disorders) | 4 (4)
Cytomegalovirus colitis (Gastrointestinal disorders) | 1 (2)
Invasive fungal infection (Infections and infestations) | 1 (1)
Acute nephrotoxicity (Renal and urinary disorders) | 1 (2)
Acute Respiratory Distress (Infections and infestations) | 1 (1)
Liver Failure (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stem Cell Transplantation in Patients With Progressive and Incurable Metastatic Solid Tumors (N=42)
Hemorrhagic cystitis (Renal and urinary disorders) | 4
Cytomegalovirus disease (Infections and infestations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-23): https://cdn.clinicaltrials.gov/large-docs/80/NCT00001880/Prot_SAP_000.pdf